CLINICAL TRIAL: NCT01820260
Title: Safety and Efficacy of Escalating Doses of Ingenol Mebutate Once Daily for Two or Three Consecutive Days When Used on Full Face, Full Balding Scalp or Approximately 250 cm2 on the Chest in Subjects With Actinic Keratosis
Brief Title: Safety and Efficacy of Ingenol Mebutate Once Daily for 2 or 3 Consecutive Days in Subjects With Actinic Keratosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LP0105-1012
Record Dates: First submitted 2013-03-25; First posted 2013-03-28 (Estimated); Results first posted 2021-05-25 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2021-05

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Intervention Model Description: Part 1 was an open-label, dose escalation. Part 2 was a randomised, double-blind, parallel group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking only for Part 2
Oversight: Data Monitoring Committee: No

ARMS (14):
- Part 1A: Ingenol mebutate gel 0.005% (Experimental): Open-label, dose escalation, 3 days treatment
  Interventions: Drug: Ingenol mebutate gel
- Part 2: Ingenol mebutate gel 0.018% for 3 days treatment (Active Comparator): Randomized, 3 days treatment
  Interventions: Drug: Ingenol mebutate gel
- Part 2: Ingenol mebutate gel 0.018% for 2 days treatment (Active Comparator): Randomized 2 days treatment
  Interventions: Drug: Ingenol mebutate gel
- Part 2: Ingenol mebutate gel 0.027% for 3 days treatment (Active Comparator): Randomized 3 days treatment
  Interventions: Drug: Ingenol mebutate gel
- Part 2: Ingenol mebutate gel 0.027% for 2 days treatment (Active Comparator): Randomized 2 days treatment
  Interventions: Drug: Ingenol mebutate gel
- Part 2: Placebo for 3 days treatment (Placebo Comparator): Randomized 3 days treatment
  Interventions: Drug: placebo
- Part 2: Placebo for 2 days treatment (Placebo Comparator): Randomized 2 days treatment
  Interventions: Drug: placebo
- Part 1A: Ingenol mebutate gel 0.008% (Experimental): Open-label, dose escalation, 3 days treatment
  Interventions: Drug: Ingenol mebutate gel
- Part 1A: Ingenol mebutate gel 0.012% (Experimental): Open-label, dose escalation, 3 days treatment
  Interventions: Drug: Ingenol mebutate gel
- Part 1A: Ingenol mebutate gel 0.027% (Experimental): Open-label, dose escalation, 3 days treatment
  Interventions: Drug: Ingenol mebutate gel
- Part 1A: Ingenol mebutate gel 0.04% (Experimental): Open-label, dose escalation, 3 days treatment
  Interventions: Drug: Ingenol mebutate gel
- Part 1B: Ingenol mebutate gel 0.06% (Experimental): Open-label, dose escalation, 2 days treatment
  Interventions: Drug: Ingenol mebutate gel
- Part 1A: Ingenol mebutate gel 0.018% (Experimental): Open-label, dose escalation, 3 days treatment
  Interventions: Drug: Ingenol mebutate gel
- Part 1B: Ingenol mebutate gel 0.04% (Experimental): Open-label, dose escalation, 2 days treatment
  Interventions: Drug: Ingenol mebutate gel

INTERVENTIONS:
Drug: Ingenol mebutate gel
  Arms: Part 1A: Ingenol mebutate gel 0.005%; Part 1A: Ingenol mebutate gel 0.008%; Part 1A: Ingenol mebutate gel 0.012%; Part 1A: Ingenol mebutate gel 0.018%; Part 1A: Ingenol mebutate gel 0.027%; Part 1A: Ingenol mebutate gel 0.04%; Part 1B: Ingenol mebutate gel 0.04%; Part 1B: Ingenol mebutate gel 0.06%; Part 2: Ingenol mebutate gel 0.018% for 2 days treatment; Part 2: Ingenol mebutate gel 0.018% for 3 days treatment; Part 2: Ingenol mebutate gel 0.027% for 2 days treatment; Part 2: Ingenol mebutate gel 0.027% for 3 days treatment
Drug: placebo
  Arms: Part 2: Placebo for 2 days treatment; Part 2: Placebo for 3 days treatment

SUMMARY:
To identify the Maximum Tolerated Dose levels of ingenol mebutate gel after once daily treatment for 2 or 3 consecutive days and to evaluate efficacy of ingenol mebutate gel in different doses after once daily treatment for 2 or 3 consecutive days compared to vehicle gel

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be competent to understand the nature of the trial and provide informed consent
* Part 1: Subjects with 5 to 20 clinically typical, visible and discrete AKs on the face Part 2: Subjects with 5 to 20 clinically typical, visible and discrete AKs on either the face, the balding scalp (the balding part of the scalp should be at least 25 cm2) or a contiguous area of approximately 250 cm2 on the chest
* Subject at least 18 years of age
* Female subjects must be of either:

  1. Non-childbearing potential, i.e. post-menopausal or have a confirmed clinical history of sterility (e.g. the subject is without a uterus) or,
  2. Childbearing potential, provided there is a confirmed negative urine pregnancy test prior to trial treatment, to rule out pregnancy
* Female subjects of childbearing potential1 must be willing to use effective contraception at trial entry and until completion

Exclusion Criteria:

* Location of the treatment area (full face, full balding scalp or chest)

  * within 5 cm of an incompletely healed wound,
  * within 10 cm of a suspected basal cell carcinoma (BCC) or squamous cell carcinoma (SCC
* Prior treatment with ingenol mebutate gel within the treatment area
* Lesions in the treatment areas that have:

  * atypical clinical appearance (e.g., hypertrophic, hyperkeratotic or cutaneous horns) and/or,
  * recalcitrant disease (e.g., did not respond to cryotherapy on two previous occasions
* History or evidence of skin conditions other than the trial indication that would interfere with the evaluation of the trial medication (e.g., eczema, unstable psoriasis, xeroderma pigmentosum)
* Use of cosmetic or therapeutic products and procedures which could interfere with the assessments of the treatment areas.
* Clinical diagnosis/history or evidence of any medical condition that would expose a subject to an undue risk of a significant AE or interfere with assessments of safety and efficacy during the course of the trial, as determined by the investigator's clinical judgment
* Any abnormal laboratory tests that are medically significant and would impact the safety of the subjects or the interpretation of the trial results, as determined by the investigator's judgment
* Anticipated need for hospitalisation or out-patient surgery during the first 15 days after the first trial medication application. Note that cosmetic/therapeutic procedures are not excluded if they fall outside of the criteria detailed in Prohibited Therapies or Medications
* Known sensitivity or allergy to any of the ingredients in ingenol mebutate gel
* Presence of acute sunburn within the treatment areas
* Current enrolment or participation in an investigational clinical trial within 30 days of entry into this trial.
* Subjects previously assigned to treatment in Part 1 or rand
* Female subjects who are breastfeeding.
* In the opinion of the investigator, the subject is unlikely to comply with the Clinical Study Protocol (e.g. alcoholism, drug dependency or psychotic state)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2013-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C. William Hanke, MD, Principal Investigator — Laser & Skin Surgery Center of Indiana
Locations (1):
- Laser & Skin Surgery Center of Inidana, Carmel, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part 1: There was 1 of the 82 subjects who withdrew before receiving any treatment but after collection of baseline characteristics. 81 subjects received treatment and all completed the trial.
  Part 2: There were 2 of the 315 randomized subjects who withdrew consent prior to any baseline characteristics being recorded (therefore they received no treatment) and are excluded from the total number of participants, full analysis set and safety analysis.
Groups:
- Part 1A: Ingenol Mebutate Gel 0.005%; Part 1A: Ingenol Mebutate Gel 0.008%; Part 1A: Ingenol Mebutate Gel 0.012%; Part 1A: Ingenol Mebutate Gel 0.018%; Part 1A: Ingenol Mebutate Gel 0.027%; Part 1A: Ingenol Mebutate Gel 0.04%: Administration on full face, once daily for 3 consecutive days
- Part 1B: Ingenol Mebutate Gel 0.06%; Part 1B: Ingenol Mebutate Gel 0.04%: Administration on full face, once daily for 2 consecutive days
- Part 2: Ingenol Mebutate Gel 0.018% for 2 Days; Part 2: Ingenol Mebutate Gel 0.027% for 2 Days: Administration on full face, full balding scalp, or approximately 250 cm² on the chest, once daily for 2 consecutive days
- Part 2: Ingenol Mebutate Gel 0.018% for 3 Days; Part 2: Ingenol Mebutate Gel 0.027% for 3 Days: Administration on full face, full balding scalp, or approximately 250 cm² on the chest, once daily for 3 consecutive days
- Part 2: Vehicle Gel (Placebo) for 2 Days: Vehicle gel administration on full face, full balding scalp, or approximately 250 cm² on the chest, once daily for 2 consecutive days
- Part 2: Vehicle Gel (Placebo) for 3 Days: Vehicle gel administration on full face, full balding scalp, or approximately 250 cm² on the chest, once daily for 3 consecutive days
Period: Phase 1 (Part 1)
Arm/Group | Part 1A: Ingenol Mebutate Gel 0.005% | Part 1A: Ingenol Mebutate Gel 0.008% | Part 1A: Ingenol Mebutate Gel 0.012% | Part 1A: Ingenol Mebutate Gel 0.018% | Part 1A: Ingenol Mebutate Gel 0.027% | Part 1A: Ingenol Mebutate Gel 0.04% | Part 1B: Ingenol Mebutate Gel 0.06% | Part 1B: Ingenol Mebutate Gel 0.04% | Part 2: Ingenol Mebutate Gel 0.018% for 2 Days | Part 2: Ingenol Mebutate Gel 0.018% for 3 Days | Part 2: Ingenol Mebutate Gel 0.027% for 2 Days | Part 2: Ingenol Mebutate Gel 0.027% for 3 Days | Part 2: Vehicle Gel (Placebo) for 2 Days | Part 2: Vehicle Gel (Placebo) for 3 Days
Started | 3 | 12 | 10 | 12 | 12 | 10 | 12 | 11 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 12 | 10 | 12 | 12 | 10 | 11 | 11 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Subject withdrew after randomization before treatment assignment | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 2 (Part 2)
Arm/Group | Part 1A: Ingenol Mebutate Gel 0.005% | Part 1A: Ingenol Mebutate Gel 0.008% | Part 1A: Ingenol Mebutate Gel 0.012% | Part 1A: Ingenol Mebutate Gel 0.018% | Part 1A: Ingenol Mebutate Gel 0.027% | Part 1A: Ingenol Mebutate Gel 0.04% | Part 1B: Ingenol Mebutate Gel 0.06% | Part 1B: Ingenol Mebutate Gel 0.04% | Part 2: Ingenol Mebutate Gel 0.018% for 2 Days | Part 2: Ingenol Mebutate Gel 0.018% for 3 Days | Part 2: Ingenol Mebutate Gel 0.027% for 2 Days | Part 2: Ingenol Mebutate Gel 0.027% for 3 Days | Part 2: Vehicle Gel (Placebo) for 2 Days | Part 2: Vehicle Gel (Placebo) for 3 Days
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 64 | 62 | 61 | 64 | 31 | 31
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 64 | 61 | 61 | 64 | 31 | 31
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: For the Safety Analysis set for Part 1 the was 1 subject out of 12 not included in the Part 1B Ingenol Mebute Gel 0.06%. This subject discontinued before receiving any trial medication. Therefore, there are only 11 subjects.
Groups:
- Part 1A: Ingenol Mebutate Gel 0.005%; Part 1A: Ingenol Mebutate Gel 0.008%; Part 1A: Ingenol Mebutate Gel 0.012%; Part 1A: Ingenol Mebutate Gel 0.018%; Part 1A: Ingenol Mebutate Gel 0.027%; Part 1A: Ingenol Mebutate Gel 0.04%: Administration on full face, once daily for 3 days
- Part 1B: Ingenol Mebutate Gel 0.04%; Part 1B: Ingenol Mebutate Gel 0.06%: Administration on full face, once daily for 2 days
- Part 2: Ingenol Mebutate Gel 0.018% for 3 Days Treatment: Administration on full face, full balding scalp, or approximately 250 cm² on the chest, once daily for 3 consecutive days
  Ingenol mebutate gel 0.018%
- Part 2: Ingenol Mebutate Gel 0.027% for 3 Days Treatment: Administration on full face, full balding scalp, or approximately 250 cm² on the chest, once daily for 3 consecutive days
  Ingenol mebutate gel 0.027%
- Part 2: Ingenol Mebutate Gel 0.018% for 2 Days Treatment: Administration on full face, full balding scalp, or approximately 250 cm² on the chest, once daily for 2 consecutive days
  Ingenol mebutate gel 0.018%
- Part 2: Ingenol Mebutate Gel 0.027% for 2 Days Treatment: Administration on full face, full balding scalp, or approximately 250 cm² on the chest, once daily for 2 consecutive days
  Ingenol mebutate gel 0.027%
- Part 2: Vehicle Gel (Placebo)for 2 Days Treatment: Vehicle gel administration on full face, full balding scalp, or approximately 250 cm² on the chest, once daily for 2 consecutive days
  Vehicle gel (placebo)
- Part 2: Vehicle Gel (Placebo) for 3 Days Treatment: Vehicle gel administration on full face, full balding scalp, or approximately 250 cm² on the chest, once daily for 3 consecutive days
  Vehicle gel (placebo)
- Total: Total of all reporting groups
Arm/Group | Part 1A: Ingenol Mebutate Gel 0.005% | Part 1A: Ingenol Mebutate Gel 0.008% | Part 1A: Ingenol Mebutate Gel 0.012% | Part 1A: Ingenol Mebutate Gel 0.018% | Part 1A: Ingenol Mebutate Gel 0.027% | Part 1A: Ingenol Mebutate Gel 0.04% | Part 1B: Ingenol Mebutate Gel 0.04% | Part 1B: Ingenol Mebutate Gel 0.06% | Part 2: Ingenol Mebutate Gel 0.018% for 3 Days Treatment | Part 2: Ingenol Mebutate Gel 0.027% for 3 Days Treatment | Part 2: Ingenol Mebutate Gel 0.018% for 2 Days Treatment | Part 2: Ingenol Mebutate Gel 0.027% for 2 Days Treatment | Part 2: Vehicle Gel (Placebo)for 2 Days Treatment | Part 2: Vehicle Gel (Placebo) for 3 Days Treatment | Total
Number analyzed (Participants) | 3 | 12 | 10 | 12 | 12 | 10 | 11 | 12 | 62 | 64 | 64 | 61 | 31 | 31 | 395
Age, Continuous [Mean (Full Range); unit: years] | 75.3 [72 to 78] | 69.6 [51 to 85] | 68.7 [48 to 81] | 67.4 [41 to 83] | 69.7 [56 to 84] | 68.0 [47 to 85] | 67.5 [57 to 83] | 71.7 [52 to 92] | 68.0 [46 to 88] | 66.3 [49 to 88] | 66.9 [47 to 91] | 66.1 [50 to 84] | 68.4 [48 to 83] | 69.0 [43 to 87] | 68.0 [41 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 2 | 1 | 2 | 1 | 5 | 20 | 15 | 8 | 15 | 3 | 5 | 79
  Male | 3 | 11 | 9 | 10 | 11 | 8 | 10 | 7 | 42 | 49 | 56 | 46 | 28 | 26 | 316
Region of Enrollment [Number; unit: participants]
  United States | 3 | 12 | 10 | 12 | 12 | 10 | 11 | 12 | 62 | 64 | 64 | 61 | 31 | 31 | 395

OUTCOME MEASURES:

1. Primary Outcome: Part 1: To Identify the Maximum Tolerated Dose (MTD) Levels After Once Daily Treatment for 2 or 3 Days
Description: Dose tolerability was measures looking at the composite score of Local Skin Responses (LSR). The MTD was defined as the highest dose level with less than 4 subjects out of 12 experiencing dose limiting toxicity (DLT).
  DLT was defined as one or more of the following three local skin LSRs:
  * Crusting Grade 4
  * Erosion/Ulceration Grade 4
  * Vesiculation/Pustulation Grade 4 or two or more of the following five LSRs:
  * Erythema Grade 4
  * Crusting Grade 3
  * Swelling Grade 4
  * Erosion/Ulceration Grade 3
  * Vesiculation/Pustulation Grade 3
  The grading is a scale of 1 to 4 (highest grade).
Time Frame: 8 days after initial treatment
Population: The composite (sum) score was obtained by summing the 6 individual LSRs
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: Ingenol Mebutate Gel 0.005% | Part 1A: Ingenol Mebutate Gel 0.008% | Part 1A: Ingenol Mebutate Gel 0.012% | Part 1A: Ingenol Mebutate Gel 0.018% | Part 1A: Ingenol Mebutate Gel 0.027% | Part 1A: Ingenol Mebutate Gel 0.04% | Part 1B: Ingenol Mebutate Gel 0.04% | Part 1B: Ingenol Mebutate Gel 0.06%
Number analyzed (Participants) | 3 | 12 | 10 | 12 | 12 | 10 | 11 | 11
Participants | 0 | 0 | 0 | 1 | 1 | 4 | 1 | 0

2. Primary Outcome: Part 2: Number of Subjects With Complete Clearance of AKs
Description: Number of subjects with complete clearance of Actinic Keratosis lesions (AKs) at week 8 after 2 or 3 consecutive days of treatment with ingenol mebutate gel on the full face, full balding scalp or approximately 250 cm² on the chest
Time Frame: 8 weeks
Measure: Number; unit: participants
Groups:
- Ingenol Mebutate Gel 0.018% for 3 Days: Administration on full face, full balding scalp, or approximately 250 cm² on the chest, once daily for 3 consecutive days
  Ingenol mebutate gel 0.018%
- Ingenol Mebutate Gel 0.018% for 2 Days: Administration on full face, full balding scalp, or approximately 250 cm² on the chest, once daily for 2 consecutive days
  Ingenol mebutate gel 0.018%
- Ingenol Mebutate Gel 0.027% for 3 Days: Administration on full face, full balding scalp, or approximately 250 cm² on the chest, once daily for 3 consecutive days
  Ingenol mebutate gel 0.027%
- Ingenol Mebutate Gel 0.027% for 2 Days: Administration on full face, full balding scalp, or approximately 250 cm² on the chest, once daily for 2 consecutive days
  Ingenol mebutate gel 0.027%
- Vehicle Gel (Placebo) for 3 Days: Vehicle gel administration on full face, full balding scalp, or approximately 250 cm² on the chest, once daily for 3 consecutive days
  Vehicle gel (placebo)
- Vehicle Gel (Placebo) for 2 Days: Vehicle gel administration on full face, full balding scalp, or approximately 250 cm² on the chest, once daily for 2 consecutive days
  Vehicle gel (placebo
Arm/Group | Ingenol Mebutate Gel 0.018% for 3 Days | Ingenol Mebutate Gel 0.018% for 2 Days | Ingenol Mebutate Gel 0.027% for 3 Days | Ingenol Mebutate Gel 0.027% for 2 Days | Vehicle Gel (Placebo) for 3 Days | Vehicle Gel (Placebo) for 2 Days
Number analyzed (Participants) | 62 | 64 | 64 | 61 | 31 | 31
participants | 15 | 19 | 25 | 13 | 1 | 0
Statistical Analysis 1: Comparison: Ingenol Mebutate Gel 0.018% for 2 Days vs Vehicle Gel (Placebo) for 2 Days; Complete clearance of AKs at Week 8 was to be analysed by log binomial regression with factors treatment group, anatomical location (face/chest or scalp) and analysis site. Due to the low numbers of subjects obtaining complete clearance in the vehicle groups,the proposed model did not converge and Fisher's exact test was used instead to compare active treatments with the respective vehicle arm; Test type: Superiority or Other; p = 0.0002, Fisher Exact — To account for multiple testing, the 4 pairwise tests with corresponding vehicle group were performed using Bonferroni method testing at a 1.25% significance level, securing that the overall significance level did not exceed 5%
Statistical Analysis 2: Comparison: Ingenol Mebutate Gel 0.027% for 2 Days vs Vehicle Gel (Placebo) for 2 Days; See comment in analysis 1; Test type: Superiority or Other; p = 0.0037, Fisher Exact — see comments in analysis 1
Statistical Analysis 3: Comparison: Ingenol Mebutate Gel 0.018% for 3 Days vs Vehicle Gel (Placebo) for 3 Days; See comments in analysis 1; Test type: Superiority or Other; p = 0.0171, Fisher Exact — See comments in analysis 1
Statistical Analysis 4: Comparison: Ingenol Mebutate Gel 0.027% for 3 Days vs Vehicle Gel (Placebo) for 3 Days; Test type: Superiority or Other; p = 0.0001, Fisher Exact

3. Secondary Outcome: Part 2: Reduction in AK Count
Description: Reduction in actinic keratosis lesion count from baseline to week 8 (percentage, adjusted for anatomical location and pooled site)
Time Frame: From baseline to Week 8
Measure: Number (95% Confidence Interval); unit: Percentage reduction
Groups:
- Ingenol Mebutate Gel 0.018% for 3 Days Treatment: Administration on full face, full balding scalp, or approximately 250 cm² on the chest, once daily for 3 consecutive days
  Ingenol mebutate gel 0.018%
- Ingenol Mebutate Gel 0.018% for 2 Days Treatment: Administration on full face, full balding scalp, or approximately 250 cm² on the chest, once daily for 2 consecutive days
  Ingenol mebutate gel 0.018%
- Ingenol Mebutate Gel 0.027% for 3 Days Treatment: Administration on full face, full balding scalp, or approximately 250 cm² on the chest, once daily for 3 consecutive days
  Ingenol mebutate gel 0.027%
- Ingenol Mebutate Gel 0.027% for 2 Days Treatment: Administration on full face, full balding scalp, or approximately 250 cm² on the chest, once daily for 2 consecutive days
  Ingenol mebutate gel 0.027%
- Vehicle Gel (Placebo) for 3 Days Treatment: Vehicle gel administration on full face, full balding scalp, or approximately 250 cm² on the chest, once daily for 3 consecutive days
  Vehicle gel (placebo)
- Vehicle Gel (Placebo)for 2 Days Treatment: Vehicle gel administration on full face, full balding scalp, or approximately 250 cm² on the chest, once daily for 2 consecutive days
  Vehicle gel (placebo)
Arm/Group | Ingenol Mebutate Gel 0.018% for 3 Days Treatment | Ingenol Mebutate Gel 0.018% for 2 Days Treatment | Ingenol Mebutate Gel 0.027% for 3 Days Treatment | Ingenol Mebutate Gel 0.027% for 2 Days Treatment | Vehicle Gel (Placebo) for 3 Days Treatment | Vehicle Gel (Placebo)for 2 Days Treatment
Number analyzed (Participants) | 62 | 64 | 64 | 61 | 31 | 31
Percentage reduction | 73.5 [66.4 to 79.1] | 70.5 [62.8 to 76.6] | 82.9 [77.6 to 86.9] | 67.7 [59.1 to 74.5] | 4.3 [-28.1 to 28.5] | 15.7 [-12.9 to 37.1]
Statistical Analysis 1: Comparison: Ingenol Mebutate Gel 0.018% for 3 Days Treatment vs Vehicle Gel (Placebo) for 3 Days Treatment; To account for multiple testing among the secondary endpoints, a hierarchical order of testing was determined, where the following evaluation was done separately for each of the four active groups: Provided the primary endpoint was significant at a 1.25% level, the comparison to vehicle in terms of reduction in AK count from baseline to week 8 was tested at a 1.25% level. Provided this test was significant, the second secondary endpoint,partial clearance, was tested(vs. vehicle) at a 1.25% level; Test type: Superiority or Other; p < 0.001, z-test
Statistical Analysis 2: Comparison: Ingenol Mebutate Gel 0.018% for 2 Days Treatment vs Vehicle Gel (Placebo)for 2 Days Treatment; See comment in analysis 1; Test type: Superiority or Other; p < 0.001, z-test
Statistical Analysis 3: Comparison: Ingenol Mebutate Gel 0.027% for 3 Days Treatment vs Vehicle Gel (Placebo) for 3 Days Treatment; See comment analysis 1; Test type: Superiority or Other; p < 0.001, z-test
Statistical Analysis 4: Comparison: Ingenol Mebutate Gel 0.027% for 2 Days Treatment vs Vehicle Gel (Placebo)for 2 Days Treatment; See comment in analysis 1; Test type: Superiority or Other; p < 0.001, z-test

4. Secondary Outcome: Part 2: Number of Subjects With Partial Clearance of AKs
Description: Partial clearance of AKs at Week 8, defined as at least 75% reduction from baseline in the number of clinically visible AKs
Time Frame: Week 8
Measure: Number; unit: percentage of participants
Arm/Group | Ingenol Mebutate Gel 0.018% for 3 Days Treatment | Ingenol Mebutate Gel 0.018% for 2 Days Treatment | Ingenol Mebutate Gel 0.027% for 3 Days Treatment | Ingenol Mebutate Gel 0.027% for 2 Days Treatment | Vehicle Gel (Placebo) for 3 Days Treatment | Vehicle Gel (Placebo)for 2 Days Treatment
Number analyzed (Participants) | 62 | 64 | 62 | 61 | 31 | 31
percentage of participants | 54.8 | 57.8 | 76.6 | 52.5 | 6.5 | 12.9
Statistical Analysis 1: Comparison: Ingenol Mebutate Gel 0.018% for 3 Days Treatment vs Vehicle Gel (Placebo) for 3 Days Treatment; Analysis of partial clearance of AK's at Week 8 was done in the same way as for the primary outcome (endpoint); Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Ingenol Mebutate Gel 0.018% for 2 Days Treatment vs Vehicle Gel (Placebo)for 2 Days Treatment; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 3: Comparison: Ingenol Mebutate Gel 0.027% for 3 Days Treatment vs Vehicle Gel (Placebo) for 3 Days Treatment; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 4: Comparison: Ingenol Mebutate Gel 0.027% for 2 Days Treatment vs Vehicle Gel (Placebo)for 2 Days Treatment; Test type: Superiority or Other; p < 0.001, Fisher Exact

ADVERSE EVENTS:
Groups:
- Part 1A: Ingenol Mebutate Gel 0.005%; Part 1A: Ingenol Mebutate Gel 0.008%; Part 1A: Ingenol Mebutate Gel 0.012%; Part 1A: Ingenol Mebutate Gel 0.018%; Part 1A: Ingenol Mebutate Gel 0.027%; Part 1A: Ingenol Mebutate Gel 0.04%; Part 1B: Ingenol Mebutate Gel 0.06%: Administration on full face, once daily 3 days
- Part 1B: Ingenol Mebutate Gel 0.04%: Administration on full face, once daily 2 days
Arm/Group | Part 1A: Ingenol Mebutate Gel 0.005% | Part 1A: Ingenol Mebutate Gel 0.008% | Part 1A: Ingenol Mebutate Gel 0.012% | Part 1A: Ingenol Mebutate Gel 0.018% | Part 1A: Ingenol Mebutate Gel 0.027% | Part 1A: Ingenol Mebutate Gel 0.04% | Part 1B: Ingenol Mebutate Gel 0.04% | Part 1B: Ingenol Mebutate Gel 0.06% | Part 2: Ingenol Mebutate Gel 0.018% for 3 Days | Part 2: Ingenol Mebutate Gel 0.018% for 2 Days | Part 2: Ingenol Mebutate Gel 0.027% for 3 Days | Part 2: Ingenol Mebutate Gel 0.027% for 2 Days | Part 2: Vehicle Gel (Placebo) for 3 Days | Part 2: Vehicle Gel (Placebo) for 2 Days
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/12 | 0/10 | 0/12 | 0/12 | 0/10 | 0/11 | 0/11 | 0/62 | 0/64 | 0/64 | 0/61 | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/12 | 0/10 | 0/12 | 0/12 | 0/10 | 0/11 | 0/11 | 0/62 | 0/64 | 0/64 | 0/61 | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 1/3 | 7/12 | 9/10 | 10/12 | 12/12 | 10/10 | 11/11 | 10/11 | 58/62 | 59/64 | 60/64 | 58/61 | 8/31 | 8/31
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1A: Ingenol Mebutate Gel 0.005% (N=3) | Part 1A: Ingenol Mebutate Gel 0.008% (N=12) | Part 1A: Ingenol Mebutate Gel 0.012% (N=10) | Part 1A: Ingenol Mebutate Gel 0.018% (N=12) | Part 1A: Ingenol Mebutate Gel 0.027% (N=12) | Part 1A: Ingenol Mebutate Gel 0.04% (N=10) | Part 1B: Ingenol Mebutate Gel 0.04% (N=11) | Part 1B: Ingenol Mebutate Gel 0.06% (N=11) | Part 2: Ingenol Mebutate Gel 0.018% for 3 Days (N=62) | Part 2: Ingenol Mebutate Gel 0.018% for 2 Days (N=64) | Part 2: Ingenol Mebutate Gel 0.027% for 3 Days (N=64) | Part 2: Ingenol Mebutate Gel 0.027% for 2 Days (N=61) | Part 2: Vehicle Gel (Placebo) for 3 Days (N=31) | Part 2: Vehicle Gel (Placebo) for 2 Days (N=31)
Application site pain (General disorders) | 0 | 5 | 8 | 8 | 12 | 9 | 11 | 9 | 56 | 56 | 60 | 57 | 2 | 4
Application site pruritus (General disorders) | 0 | 0 | 4 | 2 | 1 | 2 | 6 | 2 | 18 | 10 | 9 | 9 | 0 | 0
Application site discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 3 | 2 | 3 | 0 | 0
Application site paraesthesia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 3 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 1
Appilcation site dryness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0
Cyst rupture (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngititis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 2 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 2 | 0 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 2 | 1 | 3 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Application site reaction (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Application site oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tenderness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
oral herpes (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
upper airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No